CLINICAL TRIAL: NCT07266636
Title: Comparative Effect of Photobiomodulation and Electrical Stimulation on Facial Disability Among Bell's Palsy Patients
Brief Title: Effects of Photobiomodulation and Electrical Stimulation Among Bell's Palsy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/037 Kashaf
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Bell's Palsy
Keywords: Photobiomodulation; Electrical Muscle Stimulation; Facial Exercises
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Intervention Model Description: Group A: The participants will recieve Photobiomodulation therapy alongwith facial exercises Group B: The participants will receive Electrical Muscle Stimulation alongwith facial exercises
Who Masked: Participant, Outcomes Assessor
Masking Description: outcome assessor will be blind about participants allocation. This will ensure that their evaluations are objective and not influenced by knowledge of which treatment group participants belongs to. Participants in both groups will be masked to the treatment of the other group by scheduling their sessions at different times
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation along with facial exercises (Experimental): Group A will receive Photobiomodulation therapy alongwith facial exercises. The intervention phase will last for 5-6 weeks, with participants receiving treatment 4-5 times per week, each session lasting 30-40 minutes, under therapist supervision.
  Interventions: Radiation: Photobiomodulation alongwith facial exercise
- Electrical Muscle Stimulation alongwith facial exercises (Active Comparator): Group B will receive Electrical Muscle Stimulation therapy alongwith facial exercises. The intervention phase will last for 5-6 weeks, with participants receiving treatment 4-5 times per week, each session lasting 30-40 minutes, under therapist supervision. Group A
  Interventions: Other: Electrical Stimulation alongwith facial exercise

INTERVENTIONS:
Radiation: Photobiomodulation alongwith facial exercise — The intervention phase will last for 5-6 weeks, with participants receiving treatment 4-5 times per week, each session lasting 30-40 minutes, under therapist supervision.
  PBM therapy will be administered using a low-level laser therapy (LLLT) device, with appropriate settings (e.g., wavelength, energy density, and duration). Each session will focus on treating the affected facial regions.
  Facial Exercise will include manual therapy aimed at improving facial muscle tone, mobility, and circulation, customized for Bell's Palsy.
  Arms: Photobiomodulation along with facial exercises
Other: Electrical Stimulation alongwith facial exercise — The intervention phase will last for 5-6 weeks, with participants receiving treatment 4-5 times per week, each session lasting 30-40 minutes, under therapist supervision.
  EMS will be applied to the affected facial muscles using appropriate device settings. The therapy will focus on stimulating motor function and improving muscle tone.
  Facial Exercise will be performed as described above in Group 1 to aid in relaxation and muscle tone restoration.
  Arms: Electrical Muscle Stimulation alongwith facial exercises

SUMMARY:
Despite promising evidence supporting both photobiomodulation (PBM) and electrical stimulation (ES) in Bell's palsy rehabilitation, key gaps remain in the literature. Few studies have directly compared these modalities under standardized conditions, especially while keeping facial exercises constant across groups. Inconsistent treatment parameters such as variations in PBM wavelength or ES intensity limit the comparability and replication of existing findings. Additionally, many studies rely on subjective outcome measures and lack structured timelines for assessing facial symmetry, neuromuscular coordination, or long-term recovery, including complications like synkinesis. These limitations highlight the need for a well-controlled comparative study to determine the more effective modality when paired with consistent facial rehabilitation exercises.

DETAILED DESCRIPTION:
Bell's palsy is the most common form of lower motor neuron facial paralysis, accounting for approximately 60-75% of such cases. Although the exact cause remains unknown, it is often linked to viral infections that trigger inflammation of the facial nerve, leading to localized swelling, loss of myelin sheath, and reduced blood flow. Several factors have been identified that may increase susceptibility to the condition, including elevated blood glucose levels, poorly managed hypertension, severe pre-eclampsia, migraines, and exposure to radiation. Patients experience either partial or complete facial weakness, often accompanied by numbness, discomfort, sensitivity to sound, and changes in taste. Bell's palsy is primarily diagnosed through clinical assessment, with other potential causes being ruled out.

Among the various rehabilitative strategies, photobiomodulation (PBM) and electrical stimulation (ES) have gained significant attention. Both are non-invasive therapeutic modalities used to stimulate nerve regeneration, reduce inflammation, and promote muscle function. However, comparative studies evaluating their effectiveness in treating facial disability due to Bell's palsy remain limited. This study, therefore, aims to investigate the comparative effects of PBM and ES on facial disability in patients suffering from Bell's palsy, helping clinicians make evidence-informed decisions for optimal patient outcomes.

Physiotherapy plays a crucial role in Bell's palsy rehabilitation by targeting neuromuscular facilitation, enhancing synaptic activity, and restoring functional facial expressions. Photobiomodulation therapy, previously referred to as low-level laser therapy (LLLT), employs low-intensity lasers or light-emitting diodes (LEDs) to deliver light energy into tissues. This energy is absorbed by chromophores in cells, especially cytochrome c oxidase, triggering a cascade of biochemical events that stimulate ATP production, modulate reactive oxygen species (ROS), and reduce inflammation. These effects create a favorable environment for nerve regeneration and tissue healing.

Electrical stimulation involves applying controlled electrical currents through the skin to elicit muscle contractions. By stimulating the facial nerve or its motor endplates, ES is thought to maintain muscle tone, prevent atrophy, and potentially re-educate facial muscles through repetitive activation. Different protocols involve varying frequencies and waveforms, with surface electrodes most commonly used in clinical practice. The theoretical underpinning of both PBM and ES lies in the concept of neuroplasticity and tissue responsiveness to bioelectrical and biochemical signals. However, the optimal modality, timing, and dosage for facial nerve rehabilitation remain areas of ongoing research and debate, necessitating further empirical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with idiopathic Bell's palsy by the Physicians, moderate to severe facial muscle weakness i.e. grade III-VI on the House-Brackmann scale and duration of the condition less than 2 weeks are the inclusion criteria Exclusion Criteria
* Participants with a middle ear infection, parotid gland tumor, malignant otitis externa, tumors in the base of the lateral skull, upper motor neuron facial palsy, segmental muscle weakness, recurrent episodes of facial paralysis, polyneuropathies and Ramsay Hunt Syndrome will be excluded from the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
House-Brackmann Facial Nerve Grading System | Baseline After 6 weeks
  The HB scale categorizes facial nerve function into six grades, ranging from Grade I (normal function) to Grade VI (complete paralysis), based on assessments of symmetry at rest, degree of voluntary movement, and presence of synkinesis. It is widely used to assess the severity of facial palsy, monitor recovery after surgery or treatment, and track the progress of rehabilitation. The grading considers both resting facial appearance and movement during actions like raising the eyebrow and smiling

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Glass GE. Photobiomodulation: The Clinical Applications of Low-Level Light Therapy. Aesthet Surg J. 2021 May 18;41(6):723-738. doi: 10.1093/asj/sjab025. PMID 33471046
- [Result] Kim MH, Park SY. Population-based study and a scoping review for the epidemiology and seasonality in and effect of weather on Bell's palsy. Sci Rep. 2021 Aug 20;11(1):16941. doi: 10.1038/s41598-021-96422-4. PMID 34417505
- [Result] Rasooly D, Ioannidis JPA, Khoury MJ, Patel CJ. Family History-Wide Association Study to Identify Clinical and Environmental Risk Factors for Common Chronic Diseases. Am J Epidemiol. 2019 Aug 1;188(8):1563-1568. doi: 10.1093/aje/kwz125. PMID 31172187
- [Result] Singh A, Deshmukh P. Bell's Palsy: A Review. Cureus. 2022 Oct 11;14(10):e30186. doi: 10.7759/cureus.30186. eCollection 2022 Oct. PMID 36397921